CLINICAL TRIAL: NCT04005963
Title: The Value of PET Quantitative Analysis of Coronary Physiology in Coronary Microvascular Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XLan-S894
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: PET / CT; Coronary Microvascular Disease
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 13N-NH3 PET cardiac blood flow perfusion rest and load imaging — Immediately after the bedside injection of 13N-NH3 370 MBq, dynamic 2D collection of heart images 10 min, scanning 1 bed; , a total of 6 min), 3min bedside injection 13N?NH3 370-540 MBq immediately after the dynamic 2D collection of heart image 10 min. Both rest and load imaging are corrected for CT attenuation.
  Image reconstruction is carried out by the method of maximum expectation of an ordered subset, the dynamic image is divided into the early phase of the first 2 min and the late phase of the last 8 min, the captured image is replayed (VIP replay) of the volume image protocol and the gated data is reconstructed.

SUMMARY:
With the aging of the population and the acceleration of urbanization process, the number of cardiovascular diseases in China continues to increase, with one in five adults suffering from cardiovascular disease. The mortality rate of cardiovascular disease in China is also on the rise, and cardiovascular disease deaths are now the leading cause of death among urban and rural residents, mainly due to ischemic heart disease (IHD). Ischemic heart disease is the damage to the heart muscle caused by changes in the coronary cycle that cause an imbalance between coronary blood flow and the needs of the heart muscle.This project obtains MBF and CFR through 13N-NH3PET cardiac blood flow perfusion rest and load imaging, and explores the diagnostic value of PET imaging to CMVD. In summary, this project will obtain myocardial blood flow (MBF) and myocardial blood flow reserve (CFR) through 13N-NH3 PET cardiac blood flow perfusion rest and load imaging, explore the diagnostic value of PET imaging for CMVD, and promote the widespread application of absolute quantification of myocardial blood flow in China.

DETAILED DESCRIPTION:
With the aging of the population and the acceleration of urbanization process, the number of cardiovascular diseases in China continues to increase, with one in five adults suffering from cardiovascular disease. The mortality rate of cardiovascular disease in China is also on the rise, and cardiovascular disease deaths are now the leading cause of death among urban and rural residents, mainly due to ischemic heart disease (IHD). Ischemic heart disease is the damage to the heart muscle caused by changes in the coronary cycle that cause an imbalance between coronary blood flow and the needs of the heart muscle.

The most common cause of which is coronary arterial stenosis and blocking caused by coronary atherosclerosis, accounting for about 90% of ischemic heart disease, referred to as coronary heart disease. Coronary artery microvascular lesions .coronary microvascular disease. CMVD) is a type of coronary atherosclerosis heart disease (coronary heart disease) that refers to the clinical syndrome of labor-induced angina or myocardial ischemia caused by abnormal structure and/or dysfunction of the small and small arteries before the coronary disease under the influence of a variety of pathogenic factors. The mechanisms of myocardial ischemia include coronary atherosclerosis disease, vascular spasm disease and coronary artery microvascular dysfunction, which may overlap between three causes.

Future breakthroughs in the treatment of coronary heart disease depend on the understanding and intervention of CMVD. The incidence of CMVD is high, and studies show that more than 60% of patients with obstructive coronary heart disease co-exist CMVD coexist with CMVD, up to 67. 4% of non-obstructive coronary patients have CMVD, and the proportion of non-obstructive coronary heart disease in stable angina patients increased year by year. Studies in 11,223 patients with stable angina showed that, like obstructive coronary heart disease, non-obstructive coronary heart disease also increased the incidence of major cardiovascular adverse events in male and female patients.

Therefore, the early detection, clear diagnosis and timely treatment of CMVD is essential. At present, there are limited methods for evaluating CMVD in clinical conventional applications, including PET, transthoracic Doppler echocardiography, SPECT, CMR Traumatic techniques include selective coronary artery imaging, coronary artery doppler blood flow conduction technology, temperature dilution to measure coronary artery blood flow and CFR, microvascular resistance index. PET's greatest advantage is that it can make a variety of precise physical corrections and measure the absolute value of myocardial blood flow in rest and congestion, completely evaluate the function of the whole heart and local heart muscle, and have a higher spatial resolution than traditional SPECT; Cannot be measured repeatedly and has shortcomings such as radiation. TTDE has the advantages of non-invasive, time-saving, bedside examination, low cost and repeatable measurement, but it has high reliability only when evaluating the microvascular function of the left front drop, and the ultrasound physician must have operational experience. SPECT has high diagnostic sensitivity and negative predictive value, but it is not possible to quantify CFR, and has low spatial resolution and radiation. CMR space resolution is high, no radiation, no signal attenuation, can simultaneously detect cardiomyopathy function, tissue morphology, cardiomyopathy, cardiomyocyte and fibrosis, has gradually become a noninvasive evaluation of cardiomyopathy "gold standard", but the contrast agent in patients with renal insufficiency is prone to adverse reactions, and there are many taboo evidence. Coronary artery angiography can only show blood vessels that account for 5% of the entire coronary artery tree, with a diameter greater than l00 m, and 95% of the small blood vessels that cannot be displayed. The Coronary artery doppler blood flow guide wire measurement CFR is considered to be the "gold standard" for invasive examinations, the disadvantage of being traumatic and having trouble with operation. The temperature dilution method has a good correlation with the CFR measured by Doppler in the coronary arteries, but its measurement value will be influenced by pressure, temperature, saline injection dose and speed, salt water and blood mixing unevenly, and so on. Microvascular resistance index can specifically evaluate the microvascular function at the far end of narrow lesions, but the relationship between the measured value and cardiovascular events is not yet clear. Coronary artery microvascular function is usually assessed by detecting coronary artery blood flow reserve (coronary flow reserve, CFR) function. PET is considered the "gold standard" for noninvasive evaluation of CFR and provides absolute quantification of myocardial blood flow (MBF) and CFR. Studies have shown that CFR 2 is an independent predictor of adverse cardiovascular events, and microvascular lesions increase the risk of cardiovascular adverse events in patients after myocardial infarction. There is currently a lack of prospective clinical studies to diagnose CMVD by using PET to evaluate CFR.

This project obtains MBF and CFR through 13N-NH3PET cardiac blood flow perfusion rest and load imaging, and explores the diagnostic value of PET imaging to CMVD. In summary, this project will obtain myocardial blood flow (MBF) and myocardial blood flow reserve (CFR) through 13N-NH3 PET cardiac blood flow perfusion rest and load imaging, explore the diagnostic value of PET imaging for CMVD, and promote the widespread application of absolute quantification of myocardial blood flow in China.

ELIGIBILITY:
Inclusion Criteria:

* The patient has symptoms such as panic, chest pain, chest tightness, etc., and morphological imaging (coronary arterial CT vascular imaging (CT angiography( CTA), coronary artery imaging) is negative, or positive but does not match the symptoms;
* Recently, there are electrocardiograms, echocardiograms, cardiomyotic enzymes and other test results.

Exclusion Criteria:

* ATP or adenosine allergy;
* systolic pressure 90mmHg (1mmHg s 0.133kPa), heart rate 40 times/min, severe arrhythmia, ii degrees above room conduction block or have a history of asthma;
* acute myocardial infarction, acute myocarditis, mytalysis or endocarditis;
* acute systemic diseases or infections, uncontrolled metabolic diseases, severe lung diseases, severe liver and kidney dysfunction;
* Pregnant and lactating women.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient has symptoms such as panic, chest pain, chest tightness, etc., and morphological imaging (coronary arterial CT vascular imaging (CT angiography( CTA), coronary artery imaging) is negative, or positive but does not match the symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 13N⁃NH3,PET/CT for initial diagnosis and staging | up to 2 years
  For patient without any treatment, Initial diagnosis and staging results of 13N⁃NH3,PET/CT will be compared to pathology, clinical and follow-up result.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Xiaoli Lan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided